CLINICAL TRIAL: NCT00624481
Title: A Phase 2, 24-Week, Multicenter, Randomized, Parallel-Group, Dose-Ranging Study To Evaluate The Effect Of Teriparatide Nasal Spray On Bone Mineral Density In Postmenopausal Women With Low Bone Mineral Density
Brief Title: Study to Evaluate Effect of Intranasal Teriparatide on Bone Mineral Density in Postmenopausal Women With Low BMD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Nastech Pharmaceutical Company, Inc. (Industry)
Responsible Party: Nastech Pharmaceutical Company Inc. ( Gordon Brandt, M.D. / President ), Nastech Pharmaceutical Company Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C07-008
Record Dates: First submitted 2008-02-19; First posted 2008-02-27 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Osteopenia; Osteoporosis
Keywords: osteoporosis; osteopenia; bone mineral density; teriparatide
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Active Comparator)
  Interventions: Drug: Teriparatide
- 2 (Experimental)
  Interventions: Drug: Teriparatide Nasal Spray
- 3 (Experimental)
  Interventions: Drug: Teriparatide Nasal Spray
- 4 (Experimental)
  Interventions: Drug: Teriparatide Nasal Spray
- 5 (Experimental)
  Interventions: Drug: Teriparatide Nasal Spray

INTERVENTIONS:
Drug: Teriparatide — 20ug subcutaneous injection daily for 24 weeks
  Other Names: Forteo
  Arms: 1
Drug: Teriparatide Nasal Spray — teriparatide intranasally daily for 24 weeks
  Arms: 2
Drug: Teriparatide Nasal Spray — teriparatide intranasally daily for 24 weeks
  Arms: 3
Drug: Teriparatide Nasal Spray — teriparatide intranasally daily for 24 weeks
  Arms: 4
Drug: Teriparatide Nasal Spray — teriparatide intranasally daily for 24 weeks
  Arms: 5

SUMMARY:
This study is being conducted to compare the effect of increasing nasal teriparatide dosing on percent change in Bone Mineral Density (BMD) of the lumbar spine after 24 weeks of therapy in postmenopausal women with low bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal Female patients up to 89 years, inclusive;
* BMI ≤ 35 kg/m2, inclusive;
* In good health, determined by medical history and physical examination, as well as normal 12-lead ECG and vital signs;
* Females will be non-pregnant, non-lactating, and either post-menopausal for at least 1 year, surgically sterile (including tubal ligation, hysterectomy) for at least 3 months, until 30 days following Study Completion be willing to use an approved method of contraception;
* Have a minimum of two evaluable non-fractured lumbar vertebrae.
* Have low bone mineral density defined as having a T-score ≤ -2.0 as determined by DXA scan at either the lumbar spine (L1-L4) or total hip

Exclusion Criteria:

* Serious Medical Condition
* History of diseases which affect bone metabolism other than postmenopausal osteoporosis such as Paget's disease, any secondary causes of osteoporosis, hypoparathyroidism, or hyperparathyroidism
* Have a history of cancer within the past 5 years, except for basal cell carcinoma
* Have hypocalcemia or hypercalcemia from any cause or have a recent history of kidney stones or pre-existing hypercalciuria;
* Have used any of the mostly commonly prescribed osteoporosis medications within 3 months of starting the investigational product, or for more than 1 month at any time within 6 months prior to starting investigational product.

Max Age: 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Change in bone mineral density of the lumbar spine from baseline to 24 weeks post treatment. | 24 weeks

SECONDARY OUTCOMES:
Change in bone mineral density from baseline to 12 weeks post treatment | 12 weeks
Safety, including hypercalcemia and nasal effects | 24 weeks
Change from baseline in bone markers PINP and CTX from baseline to 4, 12 and 24 weeks post treatment | 4, 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Brandt, MD, Study Director — Nastech Pharmaceutical Company, Inc.